CLINICAL TRIAL: NCT00993356
Title: A Prospective, Randomized Trial of Preoperative Lanreotide Treatment in Acromegalic Patients With Macroadenomas
Brief Title: Preoperative Lanreotide Treatment in Acromegalic Patients With Macroadenomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: The First Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUFAH200401A
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Acromegaly
Keywords: Acromegaly; Macroadenomas; Lanreotide; Transsphenoidal neurosurgery; Preoperative
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Other): After a baseline evaluation, patients underwent transsphenoidal surgery (direct surgery group).
  Interventions: Procedure: Transsphenoidal surgery
- Group 1 (Experimental): Patients received lanreotide for 16 weeks before the surgical resection [starting with 30 mg/2 weeks i.m. and increasing to 30 mg/week i.m. at week 8, if mean GH > 5 mU/L on GH day curve (GHDC)] (GHDC: 9×30-min samples collected in the morning after an overnight fast and rest, through an indwelling catheter inserted in an arm vein and while the patient was resting).
  Interventions: Drug: Preoperative lanreotide treatment

INTERVENTIONS:
Drug: Preoperative lanreotide treatment — Patients received lanreotide for 16 weeks before the surgical resection [starting with 30 mg/2 weeks i.m. and increasing to 30 mg/week i.m. at week 8, if mean GH > 5 mU/L on GH day curve (GHDC)] (GHDC: 9×30-min samples collected in the morning after an overnight fast and rest, through an indwelling catheter inserted in an arm vein and while the patient was resting).
  Arms: Group 1
Procedure: Transsphenoidal surgery
  Arms: Group 2

SUMMARY:
Previous studies addressing preoperative somatostatin analogs (SSA) treatment and subsequent surgical cure rates are conflicting, reporting a benefit, or no difference between groups. And most reported studies were rather small and were made in retrospect, we conducted a prospective, randomized study to investigate whether 4-month preoperative lanreotide treatment would improve the surgical cure rate of newly diagnosed acromegalic patients with macroadenomas. The investigators also aimed to investigate whether there were differences in the incidence of surgical complications, and duration of neurosurgical hospital stay.

DETAILED DESCRIPTION:
Acromegaly is a rare disease, caused by a growth hormone (GH)-secreting adenoma and in even more seldom instances (about 1%) due to excessive growth hormone-releasing hormone (GHRH) secretion, usually by a carcinoid tumor of the lung or gastrointestinal tract. The incidence of acromegaly is about 3-4 per 1 million per year and the prevalence is 60-70 per 1 million, without geographical or sex differences. Clinical features of acromegaly include acral enlargement, prognathism, jaw malocclusion, arthropathy, carpal tunnel syndrome, hyperhydrosis, sleep apnea, and visceromegaly.

Transsphenoidal neurosurgery, allowing selective removal of the pituitary adenoma, is the current first treatment for acromegaly in the majority of patients. Its effects on GH and insulin-like growth factor I (IGF-I) secretion are rapid and operations have a low morbidity and very low mortality. However, surgery for macroadenomas causing acromegaly has a much lower surgical success rate than that for microadenomas. In experienced hands, microadenomas can be expected to be cured in around 90%, whereas with macroadenomas the figure is around 50%. This is particularly the case with tumours that extend into the cavernous sinus where surgical success is < 50%. Medical treatment of acromegaly with somatostatin analogs (SSAs) can lead to normalized GH and IGF-I levels and relief of symptoms. SSA treatment may cause shrinkage of GH-secreting pituitary adenomas. Theoretically, this could improve the likelihood of a radical resection, particularly in macroadenomas. Furthermore, it has been suggested that SSA treatment softens the tumor parenchyma and thereby facilitates tumor removal. Finally, it has been reported that SSA pretreatment leads to a shortening of postoperative hospital stay.

Previous studies addressing preoperative SSA treatment and subsequent surgical cure rates are conflicting, reporting a benefit, or no difference between groups. And most reported studies were rather small and were made in retrospect, we conducted a prospective, randomized study to investigate whether 4-month preoperative lanreotide treatment would improve the surgical cure rate of newly diagnosed acromegalic patients with macroadenomas. We also aimed to investigate whether there were differences in the incidence of surgical complications, and duration of neurosurgical hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed acromegaly due to GH-secreting macro-adenomas.
* newly diagnosed, previously untreated patients with GH nadir more than 2.5 μg/L during a standard 75-g, 2-h oral glucose tolerance test (OGTT)
* pituitary macroadenomas (maximum diameter >1 cm) verified by a pituitary magnetic resonance imaging (MRI) scan
* age between 18 and 80 yr.

Exclusion Criteria:

* immediate surgery indicated by clinical criteria
* pregnancy
* contraindications to MRI scan
* patients judged not suitable to participate in the study for other reasons such as personality disorders and alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2004-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Cure rate at evaluation 4 months postoperatively | every 4 weeks

SECONDARY OUTCOMES:
Postoperative hospital stay duration | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hai-jun Wang, MD, Study Director — Department of Neurosurgery, The First Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Department of Neurosurgery, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Mao ZG, He DS, Zhou J, Yao B, Xiao WW, Chen CH, Zhu YH, Wang HJ. Differential expression of microRNAs in GH-secreting pituitary adenomas. Diagn Pathol. 2010 Dec 7;5:79. doi: 10.1186/1746-1596-5-79. PMID 21138567
- [Derived] Mao ZG, Zhu YH, Tang HL, Wang DY, Zhou J, He DS, Lan H, Luo BN, Wang HJ. Preoperative lanreotide treatment in acromegalic patients with macroadenomas increases short-term postoperative cure rates: a prospective, randomised trial. Eur J Endocrinol. 2010 Apr;162(4):661-6. doi: 10.1530/EJE-09-0908. Epub 2010 Jan 8. PMID 20061334